CLINICAL TRIAL: NCT05175274
Title: Colchicine Use for Primary Prevention in People at High Risk of Coronary Artery Disease
Brief Title: Colchicine Use for Primary Prevention of Coronary Artery Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Collaborators: Qingdao Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Col-CH
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; primary prevention; adverse events
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): colchicine 0.5mg every 24 hours for 3 years
  Interventions: Drug: Colchicine
- Control Group (Placebo Comparator): 1 placebo tablet every 24 hours for 3 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5mg/tablet
  Arms: Intervention Group
Drug: Placebo — matching placebo
  Arms: Control Group

SUMMARY:
Colchicine has been widely used as an anti-gout medicine in the past decades. Some recent clinical trials have proved that low-dose colchicine can be used as a secondary prevention drug for coronary artery disease because of its anti-inflammatory mechanism. However, the effect on primary prevention has not been observed sufficiently. The objective of this study is to determine whether colchicine reduces the incidence of CAD in patients and its safety for long-term use.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who have at least 3 risk factors for CAD. 2. GFR>90mmol/L. 3 People are within 40-70 years old.4. Patients are not pre-diagnosed with CAD, which is defined by negative results of CT coronary angiography.

Exclusion Criteria:

1. Patients with any pre-existing diagnosis of coronary artery disease.2.Other cardiovascular diseases such as peripheral vascular disease, congestive heart failure and cardiomyopathy.3.Cerebrovascular diseases such as cerebral thrombosis and cerebral hemorrhage. 4.Currently on treatment with colchicine.5.Patients who are known to be allergic to colchicine.6 Chronic symptomatic heart failure within the last year and known reduced ejection fraction (LVEF≤40 %), documented before recruitment.7.Severe hepatic impairment (Child-Pugh class C) at the time of inclusion into the trial.8.Any other non cardiovascular diseases, such as active malignancy requiring treatment at the time of screening or with a life expectancy of fewer than two years based on the investigator´s clinical judgment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6792 (Estimated)
Dates: Start 2022-12-06 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of CAD | 3 years
  Collect the incidence of CAD during the follow-up time. CAD is defined with the positive stress test, ST depression in ECG with typical symptoms of myocardial ischemia, and progression to myocardial infarction. To further detect patients with occult CAD, the rest of the asymptomatic patients will be subjected to CT coronary angiography, in which CAD is defined with over 50% diameter stenosis in a major coronary artery.
Occurrence of adverse events in both groups | 3 years
  Collect the occurrence of adverse events in both groups during the drug use.Adverse events include gastrointestinal, liver, hematology, muscle, neurology, other sensory, infectious and death.

SECONDARY OUTCOMES:
MACE events | 3 years
  To assess the occurence of myocardial infarction, stroke and death from cardiovascular causes during the follow-up time.

CONTACTS AND LOCATIONS:
Locations (1):
- Mengmei Li, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No